CLINICAL TRIAL: NCT05279638
Title: Evaluation of ATG5 as Aserum Marker of Autophgy in Psoriasis Vulgaris Patients
Brief Title: ATG5 as a Serum Marker of Autophagy in Psoriatic Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ayatallah Hamdy Abdelrahim, Resident physician, Sohag University
Other Study IDs: Soh-Med-22-02-03
Record Dates: First submitted 2022-02-23; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Psoriasis Vulgaris; Autophagy
Keywords: serum marker; ATG5

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- psoriasis vulgaris patients: psoriasis vulgaris patients , both sex , 18,55 years old
  Interventions: Diagnostic Test: serum ATG5
- healthy participants
  Interventions: Diagnostic Test: serum ATG5

INTERVENTIONS:
Diagnostic Test: serum ATG5 — This kit is used to assay the Autophagy protein 5(ATG5) in the sample of human's serum, blood plasma, and other related tissue Liquid
  Other Names: human autophgy protien 5 ELISA kit

SUMMARY:
it will be of interest to know the ATG 5 as a serum marker of autophagy in serum of psoriasis vulgairs patients and explore its relationship with psoriasis severity.

ELIGIBILITY:
Inclusion Criteria:

Psoriasis vulgaris of both sex, age 18-55 years

Exclusion Criteria:

i. Patients with other types of psoriasis ii. Pregnant or lactating women iii. patients with hepatic or renal diseases iv. patients receive any systemic treatment in last 3 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with psoriasis vulgaris and healthy participatins
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
serum level of ATG5 in psoriatic patients | Within 6 months
  evaluation of serum ATG5 in psoriasis vulgaris patients by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided